CLINICAL TRIAL: NCT06764420
Title: Effect of Arginine and Glutamine on Radiation-induced Oral Mucositis: a Trible Blinded Randomized Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma ElSayed, assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: (21)/7-2024
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Radiation Mucositis; Head and Neck Cancer
Keywords: arginine; glutamine; HNC; Mucositis; Radiation
MeSH Terms: conditions — Head and Neck Neoplasms; Mucositis | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): This group includes twenty patients receiving a combined oral suspension of 5 grams of arginine and 5 grams of glutamine dissolved in cold water. The suspension is taken 30 minutes before meals, three times per day, through the swish and swallow technique throughout the radiotherapy period. This group aims to evaluate the effectiveness of the combined treatment in managing radiation-induced mucositis.
  Interventions: Dietary Supplement: Arginine and Glutamine Oral Suspension
- Control Group (Active Comparator): This group includes twenty patients receiving an oral suspension of 5 grams of glutamine dissolved in cold water. The suspension is taken 30 minutes before meals, three times per day, through the swish and swallow technique throughout the radiotherapy period. This group serves as a control to compare the efficacy of glutamine alone with the combined treatment in managing radiation-induced mucositis. General measures and analgesic drugs according to the WHO scale are also provided.
  Interventions: Dietary Supplement: Glutamine Oral Suspension

INTERVENTIONS:
Dietary Supplement: Glutamine Oral Suspension — Participants in this group will receive an oral suspension containing 5 grams of glutamine dissolved in cold water. This solution is administered 30 minutes before meals, three times per day, using the swish and swallow technique throughout the radiotherapy period. This control intervention serves to compare the effects of glutamine alone with the combined arginine and glutamine treatment. In addition to the glutamine suspension, patients in this group will receive general measures and analgesic drugs according to the WHO scale to manage symptoms of mucositis.
  Arms: Control Group
Dietary Supplement: Arginine and Glutamine Oral Suspension — Participants in this group will receive an oral suspension containing 5 grams of arginine and 5 grams of glutamine dissolved in cold water. This solution is administered 30 minutes before meals, three times per day, using the swish and swallow technique throughout the radiotherapy period. The swish and swallow technique involves patients swishing the solution around the oral mucosa to ensure even distribution before swallowing. This intervention aims to evaluate the combined effect of arginine and glutamine on reducing the severity of radiation-induced mucositis, improving mucosal healing, and providing symptomatic relief.
  Arms: Intervention Group

SUMMARY:
Oral Mucositis (OM) is a painful inflammation and ulceration of the oral mucosa, often resulting from cancer treatments like chemotherapy and radiation therapy, particularly in head and neck cancer patients. This condition is highly prevalent, affecting up to 40% of patients undergoing conventional chemotherapy, 80% of those receiving high-dose chemotherapy before hematopoietic stem cell transplantation, and nearly all patients undergoing radiation therapy for head and neck cancers.

OM develops in four phases: inflammatory/vascular, epithelial, ulcerative/bacteriological, and wound healing. The initial phase involves damage to DNA and basal epithelial cells due to free radicals and reactive oxygen species (ROS) produced by treatments. This damage leads to a cascade of inflammatory reactions, resulting in visible lesions and bacterial colonization in the subsequent stages.

Glutamine, an amino acid abundant in human blood, plays a crucial role in cellular repair, immune function, and muscle maintenance. It is a preferred energy source for lymphocytes and the gastrointestinal tract, aiding in mucosal healing and resistance to infections. Studies suggest that glutamine supplementation can reduce the toxic effects of radiation on the GI tract and improve mucosal healing by supporting immune cells and reducing inflammation.

L-arginine, another amino acid, contributes to protein synthesis, nitric oxide production, and regulation of various physiological functions. It has been shown to decrease intestinal inflammation and oxidative stress, promoting mucosal immune homeostasis. L-arginine administration has demonstrated beneficial effects in reducing intestinal injury and inflammation in experimental models.

The study proposes evaluating the combined effect of arginine and glutamine on radiation-induced mucositis in head and neck cancer patients. The primary objective is to assess the clinical efficacy of an oral suspension of these amino acids using the WHO Oral Toxicity Scale. Secondary objectives include evaluating pain and mucositis severity using assessment scales.

The hypothesis is that arginine and glutamine supplementation may reduce mucositis severity and improve clinical outcomes, potentially leading to better nutritional status, enhanced survival, and reduced complications in cancer patients.

This study aims to fill the gap in existing research by investigating the synergistic effects of these amino acids in managing radiation-induced mucositis.

DETAILED DESCRIPTION:
Oral Mucositis (OM) refers to inflammation and ulceration of the oral mucosa as a side-effect of cancer therapy. OM and esophagitis can occur secondary to systemic chemotherapy for cancer, high-dose chemotherapy as a hematopoietic transplant preparative regimen or due to radiation therapy (RT) for head and neck (H&N) cancer or if the oropharynx or esophagus is in field during and after radiation of bone metastases. OM is a common problem and occurs in about 20-40% of patients receiving conventional chemotherapy for solid tumors, about 80% of patients receiving high dose chemotherapy prior to a hematopoietic stem cell transplantation (HSCT) and almost all patients receiving RT for H&N cancer. Ulcerative OM and esophagitis are extremely painful, with many patients needing systemic opioids such as morphine or fentanyl for pain management.[1] Oral mucositis is an acute mucosal inflammation that starts as redness and progresses to an increased ulceration and pseudo membrane formation, which represent a temporary barrier until cellular repair promotes healing. The impaired mucosal tissue often permits bacteria and fungi to penetrate into damaged mucosa and cause infections.[2] Mucositis is divided into 4 phases: an initial inflammatory/ vascular phase, an epithelial phase, an ulcerative/bacteriological phase, and a wound healing phase.[3] In the initial stage, irradiation or chemotherapy, by producing free radicals and Reactive oxygen species (ROS), harmfully influences cells and strands of DNA in the basal epithelium and the submucosa and leads to lesions. ROS also activate transcription factors and leads to cell destruction in later stages. In the next stage, not only ROS but also damaged cells and DNA start a cascade of reactions. During these reactions, proinflammatory cytokines produce and lead to lesions and basal cell apoptosis. These products have a positive reaction as well, and strengthen the lesions. In this stage, the tissue appears to be normal, with only with slight erythema. In the third stage, painful lesions appear and are colonized by bacteria. Bacterial colonization can lead to the release of new pro-inflammatory cytokines. After stopping cancer treatment, oral mucositis vanishes little by little. In the healing process, symptoms decrease and the mucosa become normal, but outstanding neovascularization remains. This tissue is easily broken and it is susceptible to chemotherapy and/or radiotherapy in future periods of cancer treatments.[4]

. This diversity in scoring systems for Oral Mucositis may lead to controversies among studies. The most widely used measurements for oral mucositis are the World Health Organization(WHO) and Radiation Therapy Oncology Group (RTOG) scales as below.

Also, the Oral Mucositis Assessment Scale, and a Visual Analog Pain Scale (patient reporting scale of 0-10) are used for grading of mucositis. Mucosal changes like redness, ulceration with functional outcomes such as inability to eat and pain have been assessed in these scales. Based on clinical examination, 4 distinct grades can be determined for mucositis from 0 to 4 scores. Higher grades of mucositis (grade 3-4) are associated with loss of taste, hemorrhage, decreased intake of food and fluids, ulceration, pain, loss of voice, and low quality of life.[5] Glutamine is an L-alpha-amino acid. It is the most abundant free amino acid in human blood. Glutamine is needed for several functions in the body including for the synthesis of proteins as well as an energy source. Glutamine can be synthesized by the body and can also be obtained from the diet if needed.[6] Glutamine is an important nitrogen donor in intracellular metabolism and in the maintenance of intestinal tract, immune cells, and muscle.[7] Weight loss in cancer patients is common, but sarcopenia (loss of muscle mass) is associated with increased complications and significantly worse survival.[8] Glutamine is a preferred fuel for both lymphocytes and gastrointestinal (GI) tract [9], thus it plays an important role in helping to defend against infections and to assist mucosa in being a barrier against infection.

Glutamine has a central role in intracellular metabolism and acts as a nitrogen shuttle between muscle and other tissues; it is at a high and relatively stable concentration in plasma and red blood cells and at a much higher concentration in muscle compared to other amino acids.[10] Since plasma glutamine concentrations are only minimally affected over time by either glutamine ingestion or infusion, muscle can be considered as a "bank" and the liver can be considered as the "banker".[8] Neutrophils, macrophages, and lymphocytes are needed for mucosal barrier immune defenses. Since glutamine is fuel for leukocytes, topical/oral/enteral glutamine may contribute to mucosal healing by not only a direct effect on mucosal epithelial cells, but also by improvement in host mucosal immune function and ability to resist microbial invasion.[7] Interestingly, resilience of lymphocyte recovery, as measured by absolute lymphocyte count (ALC) after the very first cycle of chemotherapy, has been associated with a better prognosis in a variety of malignancies including acute lymphoblastic leukemia as well as tumors such as osteosarcoma, Ewing sarcoma, and rhabdomyosarcoma . It is possible that better nutrition, with amino acids including glutamine as fuel for lymphocytes, could contribute to ALC recovery and/or resilience. Animal models and human studies have shown glutamine supplementation improves the ability to resist the toxic effects of radiation to the GI tract.[6] Detoxification and resilience to free radical damage by chemotherapy (e.g., doxorubicin or cyclophosphamide) and/or radiation of normal tissues and tumors can involve the antioxidant glutathione. Since glutamine is a substrate for glutathione synthesis, adequate mucosal cell glutamine may contribute towards improved healing after chemotherapy and radiation damage [11] as well as, interestingly, the simultaneous inhibition of glutathione levels in tumors, too.[12] Furthermore, decreased inflammatory cytokines in normal cells and increased pro-apoptosis proteins in cancer cells were observed with glutamine + disaccharide supplementation. Thus, glutamine can contribute to selective improvement in host cell resilience, less inflammation, and decreased ability of tumors to detoxify chemotherapy or resist radiation, i.e. an improved therapeutic index of the anti-cancer therapy.[13] Glutamine can be administrated by three common routes: parental, oral and topical through swishing. Topical oral swish and swallow glutamine has potential to ameliorate not only OM, but also esophagitis and enteritis after cancer chemotherapy and radiation. A small amino acid intervention may make a difference and possibly contribute to better overall nutritional status, improved survival with fewer complications, and ultimately less sarcopenia and lymphopenia.[6] L-arginine (2-Amino-5-guanidinovaleric acid-Arg) is an endogenous amino acid, which is mainly formed in the urea cycle. It is involved in synthesis of proteins, urea, creatine, prolamines (purtescin, spermine, spermidine), proline and nitric oxide (NO). The end products of arginine metabolism are NO, glutamate and prolamins that have various regulatory functions in the body.[14] L-arginine is considered as a conditionally essential amino acid, which is mainly catalyzes by nitric oxide synthase (NOS), arginine decarboxylase and arginase (ARG) and arginase for synthesis of protein and several bioactive molecules such as nitric oxide (NO), proline, creatine, and polyamines.[15] Recently, there is an increasing emphasis on the improvement of the physiological functions of arginine, such as attenuating intestinal inflammation and oxidative stress.[16] Previous studies demonstrated that L-arginine administration in animals and humans with intestinal diseases can decrease intestinal injury, reduce oxidative stress and inflammation and restore mucosal immune homeostasis. Coburn et al., have reported that L-arginine administration could decreased intestinal inflammation in murine models of dextran sulfate sodium (DSS)-induced colitis, an experimental model of IBD.[17] L-arginine also showed an inhibitory effect on IL-1β-mediated NF-κB-activation in Caco-2 cells[18]. In addition, Zhang et al., demonstrated that L-arginine protected ovine intestinal epithelial cells from LPS-induced apoptosis through attenuating oxidative stress.[19] However, the precise molecular mechanism of L-arginine alleviated inflammatory response as well as decreased oxidative injury induced by LPS still remains unexplored. L-arginine serves as a degradation substrate for several enzymes in the cells, such as Arg-1. Several studies have demonstrated that Arg-1 exhibited an anti-inflammatory effect and played a beneficial role in inflammatory disease[20].

To the best of our knowledge, there are no published studies regarding using blend of arginine and glutamine in treatment of radiotherapy induced oral mucositis So regarding the forementioned properties of glutamine and arginine, we hypothized that use of arginine and glutamine could affect severity of mucositis and.

The purpose of this study is to evaluate the influence of arginine and glutamine in treatment of radiation induced mucositis in head and neck cancer patients.

Aim of the study

This randomized clinical and biochemical study will be carried out to evaluate the efficacy of locally and orally delivered arginine and glutamine in management of radiation-induced mucositis in patients with head and neck cancer.

The study will be conducted to assess:

Primary objective:

Effect of arginine and glutamine oral suspension in management of radiation induced mucositis clinically with WHO Oral Toxicity Scale Grading of Oral Mucositis.

Secondary objective:

Effect of arginine and glutamine in oral mucositis assessment score and pain visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

Confirmed histologic diagnosis of H&N malignancy.

Undergoing non-palliative radiotherapy in the oral cavity.

Receiving radiation therapy with IMRT or 3D techniques. Received 50-70 Gy of total radiation at 2 Gy/fraction daily, 5 fractions/week. Concurrent chemotherapy with radiotherapy. Presence of Oral Mucositis. Age 20-70 years. Willingness to participate and complete study assessments.

V. Exclusion Criteria:

Confirmed or medically treated diabetes mellitus. Radiotherapy within the last 6 months. Vulnerable patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
World Health Organization (WHO) Oral Toxicity Scale for grading oral mucositis. | Baseline (before the start of radiotherapy), second week of radiotherapy, seventh week of radiotherapy, and three months after the completion of radiotherapy.
  World Health Organization (WHO) Oral Toxicity Scale for grading oral mucositis. description? The World Health Organization (WHO) Oral Toxicity Scale is a standardized tool used to grade the severity of oral mucositis, which is a common side effect of cancer treatments like chemotherapy and radiotherapy. The scale helps clinicians assess and document the extent of mucositis in patients, ensuring consistent reporting and comparison across studies.
  Grade 0 No mucositis; normal oral mucosa. Grade 1 Soreness and erythema (redness) but no ulcers. Grade 2 Erythema and ulcers present, but the patient can still tolerate a solid diet.
  Grade 3 Ulcers are present, and the patient can only tolerate a liquid diet. Grade 4 Ulcers are present, and the patient cannot tolerate any oral intake (solids or liquids)

SECONDARY OUTCOMES:
Oral Mucositis Assessment Scale (OMAS) Score | Baseline (before the start of radiotherapy), second week of radiotherapy, seventh week of radiotherapy, and three months after the completion of radiotherapy.
  The Oral Mucositis Assessment Scale (OMAS) is a tool to measure the severity of oral mucositis by assessing erythema and ulcerations/pseudomembrane formation across nine intra-oral sites.
  Erythema:
  Score 0: No erythema.
  Score 1: Mild/moderate erythema (increased mucosa color intensity).
  Score 2: Severe erythema (mucosa color like fresh blood).
  Ulcerations/Pseudomembrane Formation:
  Score 0: No lesion.
  Score 1: Lesions < 1 cm².
  Score 2: Lesions 1 cm² to 3 cm².
  Score 3: Lesions > 3 cm².
  OMAS scores are calculated by summing erythema and ulceration subscores at each site. Erythema scores range from 0 to 18, and ulceration scores range from 0 to 27. The total OMAS score is averaged across affected sites, providing an overall assessment of mucositis severity.

OTHER OUTCOMES:
Pain Visual Analog Scale (VAS) | Baseline (before the start of radiotherapy), second week of radiotherapy, seventh week of radiotherapy, and three months after the completion of radiotherapy.
  Assessment of the intensity of pain associated with oral mucositis using the Visual Analog Scale (VAS), where patients rate their pain on a scale from 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Maher Teaching Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hassanein FEA, Mikhail C, Elkot S, Abou-Bakr A. L-arginine vs. L-glutamine oral suspensions for radiation-induced oral mucositis: a triple-blind randomized trial. J Cancer Res Clin Oncol. 2025 Jul 3;151(7):198. doi: 10.1007/s00432-025-06213-x. PMID 40603739